CLINICAL TRIAL: NCT00900653
Title: Low Dose Estriol With Lactobacilli (Gynoflor) Treatment for Preventing Recurrent Urinary Tract Infection in Postmenopausal Women: A Randomized, Open, Parallel-Group Study
Brief Title: Low Dose Estriol With Lactobacilli Treatment for Preventing Recurrent Urinary Tract Infection in Postmenopausal Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yonsei University (Other)
Responsible Party: Jun Yong Choi, Yonsei University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2009-0022
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Urinary Tract Infections
Keywords: urinary tract infections; postmenopause; lactobacillus; estriol
MeSH Terms: conditions — Urinary Tract Infections | interventions — Estriol; Lacteol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gynoflor (Experimental)
  Interventions: Drug: Gynoflor E (low dose estriol with lactobacillus)
- Control (No Intervention)

INTERVENTIONS:
Drug: Gynoflor E (low dose estriol with lactobacillus) — The medication, in the form of one vaginal tablet, is administered in the evenings for 18 days
  Other Names: Gynoflor E vaginal tablet
  Arms: Gynoflor

SUMMARY:
Recurrent urinary tract infections (UTI) are a problem for postmenopausal women. The aim of this trial is to evaluate the effectiveness of lactobacilli in combination with low dose estriol for preventing recurrent urinary tract infections in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman
* History of urinary tract infection
* Agree to abstain from self-medication with antibiotics for UTI symptoms
* Agree to abstain from the use of any other intra-vaginal product
* Capable of providing informed consent

Exclusion Criteria:

* Ovarian cancer, cervical cancer, breast cancer
* Estrogen treatment within last 2 years
* Vaginal bleeding
* Antibiotic therapy fewer than three days prior to randomization visit
* Known congenital urologic or gynecologic abnormalities
* Indwelling urinary catheter
* Thromboembolic disease
* Uncompensated liver disease
* Immunosuppressive drug within 60 days

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of urinary tract infection | 6 months

SECONDARY OUTCOMES:
vaginal pH | 6 months
lactobacillus colonization | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea